CLINICAL TRIAL: NCT02656823
Title: Implant-fixed Restorations With Short Implants in the Edentulous Maxilla - A Clinical Investigation Over a 5-year Follow-up Period
Brief Title: Implant-fixed Restorations With ANKYLOS 6.6 mm Implants in the Edentulous Maxilla - A 5-year Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-AN-14-001
Record Dates: First submitted 2015-12-15; First posted 2016-01-15 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Edentulous Maxilla
Keywords: ANKYLOS; Simplant; maxilla; edentulous; short implants
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- ANKYLOS C/X Implant A 6.6 (Experimental): ANKYLOS C/X Implant A 6.6 mm
  Interventions: Device: ANKYLOS C/X implant A 6.6

INTERVENTIONS:
Device: ANKYLOS C/X implant A 6.6 — Treatment with six (6) 6.6 mm implants and a bridge to restore chewing function of an edentulous maxilla.

SUMMARY:
Study to assess the performance of six short implants (ANKYLOS C/X 6.6 mm) in the edentulous maxilla supporting fixed full-arch bridges after 5 years in function.

DETAILED DESCRIPTION:
Study to assess the performance of six short implants (ANKYLOS C/X 6.6 mm) in the edentulous maxilla supporting fixed full-arch bridges after 5 years in function. The primary objective was to evaluate implant survival.

ELIGIBILITY:
INCLUSION CRITERIA

For inclusion in the study subjects had to meet all of the following criteria:

1. Aged 18-80 years at inclusion.
2. Signed informed consent.
3. In need of full-arch restoration of the maxilla.

   The following should be considered at inclusion but should be fulfilled at Implant Placement (Visit 3):
4. Maxilla: totally edentulous, fulfilling all of the following criteria:

   1. History of edentulism: ≥ 6 months and,
   2. Minimum bone height: ≥ 7 mm and,
   3. Minimum bone width: ≥ 5.5 mm.
5. Mandible: antagonistic natural dentition or tooth/implant borne rehabilitation which can be used to create a stable occlusal fit with the new full-arch restoration of the upper jaw.

EXCLUSION CRITERIA

Any of the following was regarded as a criterion for exclusion from the study:

1. Unlikely to be able to comply with study procedures according to Investigator's judgement.
2. History of bone augmentation in the maxilla within 6 months prior to surgery.
3. Uncontrolled pathologic processes in the oral cavity.
4. Bruxism.
5. Smoking >10 cigarettes per day.
6. Present alcohol or drug abuse.
7. History of radiation therapy in head and neck region.
8. History of chemotherapy within 5 years prior to surgery.
9. Condition that would compromise post-operative tissue healing or osseointegration.
10. Bisphosphonates or any other medication that would compromise post-operative healing or osseointegration.
11. Known pregnancy at time of inclusion.
12. Current or former participation in a clinical study that may interfere with the present study.
13. Involvement in the planning and conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Weigl, Principal Investigator — J. W. Goethe-Universität, Frankfurt
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implant
Groups:
- ANKYLOS C/X Implant A 6.6: Subjects treated with ANKYLOS C/X Implant A 6.6 mm.
Period: Overall Study
Arm/Group | ANKYLOS C/X Implant A 6.6
Started (Implants placed at implant placement visit (IPV), Visit 3.) | 12; 72 Implant
Permanent Restoration (PR), Visit 8 | 11; 62 Implant
Completed | 7; 41 Implant
Not Completed | 5; 31 Implant
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 12 subjects received implants in the clinical investigation.
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: Any implant that is removed after implant placement will be considered failure, whatever reason for removal. Implant survival will be evaluated clinically and radiographically by counting the number of remaining implants.
Time Frame: At Visit 14, 5 years after permanent restoration (PR).
Population: Intention to treat.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 12
Number analyzed (Implants) | 60
Implants
  Implants confirmed as survived | 41
  Implants confirmed to be failures | 19

2. Secondary Outcome: Implant Stability
Description: Implant stability was evaluated clinically/manually by the investigator at implant placement visit (this initial manual check is called primary stability), and again at the abutment surgery visit. The stability evaluation was recorded as yes/no, yes = judged by the investigator to be stable, or no = judged by the investigator to be unstable. Stability was assessed at implant placement (IP) (Visit 3), and at Abutment Surgery and Impression (Visit 5, at 13 weeks after IP).
Time Frame: At implant placement (IP) (Visit 3), and at Abutment surgery and Impression (Visit 5, at 13 weeks after IP).
Population: Intention to treat
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 12
Number analyzed (Implants) | 72
Implants
  Implant stability at Visit 3: No | 35
  Implant stability at Visit 3: Yes | 37
  Implant stability at Visit 5: No | 5
  Implant stability at Visit 5: Yes | 67

3. Secondary Outcome: Mean Marginal Bone Level (MBL) at Subject's Tissue Level
Description: The mean Marginal Bone Level (MBL) on subject level. Bone level response will be evaluated from intra-oral radiographs. The radiographs will be sent for central evaluation to a radiologist who is independent from the investigational group and the Sponsor. The radiologist will measure and record the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. The reference point is defined as the implant shoulder.
Time Frame: At permanent restoration (PR) (Visit 8, at 17 weeks after IP), and at 1-year after PR (Visit 10), at 3-years after PR (Visit 12), and at 5-years after PR (Visit 14).
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
millimeters (mm)
  Permanent restoration (Visit 8) | 1.43 (0.70)
  1-year post permanent restoration (Visit 10) | 1.44 (0.84)
  3-years post permanent restoration (Visit 12): number analyzed (Participants) | 8
  3-years post permanent restoration (Visit 12) | 1.20 (0.74)
  5-years post permanent restoration (Visit 14): number analyzed (Participants) | 7
  5-years post permanent restoration (Visit 14) | 1.17 (0.71)

4. Secondary Outcome: Mean Marginal Bone Level (MBL) on Implant Level.
Description: The mean Marginal Bone Level (MBL) on implant level. Bone level response will be evaluated from intra-oral radiographs. The radiographs will be sent for central evaluation to a radiologist who is independent from the investigational group and the Sponsor. The radiologist will measure and record the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. The reference point is defined as the implant shoulder.
Time Frame: as for outcome 3
Population: Intention to treat group. 2 implants missing from the analysis at Visit 14 (5-year follow-up).
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: implants
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
Number analyzed (implants) | 62
millimeters (mm)
  Permanent restoration (Visit 8) | 1.41 (1.13)
  1-year post permanent restoration (Visit 10): number analyzed (implants) | 60
  1-year post permanent restoration (Visit 10) | 1.42 (1.25)
  3-years post permanent restoration (Visit 12): number analyzed (Participants) | 8
  3-years post permanent restoration (Visit 12): number analyzed (implants) | 44
  3-years post permanent restoration (Visit 12) | 1.21 (1.36)
  5-years post permanent restoration (Visit 14): number analyzed (Participants) | 7
  5-years post permanent restoration (Visit 14): number analyzed (implants) | 39
  5-years post permanent restoration (Visit 14) | 1.17 (1.29)

5. Secondary Outcome: Mean Probing Pocket Depth (PPD) at Subject Level.
Description: PPD was measured as the distance from the mucosal margin to the bottom of the probeable pocket in mm.
Time Frame: At permanent restoration (PR) (Visit 8, at 17 weeks after IP), and at 6-months after PR (Visit 9), at 1-year after PR (Visit 10), at 2-years after PR (Visit 11), at 3-years after PR (Visit 12), and at 5-years after PR (Visit 14).
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
millimeter (mm)
  Permanent restoration (Visit 8) | 3.4 (0.4)
  6-months post permanent restoration (Visit 9) | 3.5 (4.7)
  1-year post permanent restoration (Visit 10) | 4.1 (4.7)
  2-years post permanent restoration (Visit 11): number analyzed (Participants) | 10
  2-years post permanent restoration (Visit 11) | 3.4 (4.4)
  3-years post permanent restoration (Visit 12): number analyzed (Participants) | 8
  3-years post permanent restoration (Visit 12) | 3.9 (4.9)
  5-years post permanent restoration (Visit 14): number analyzed (Participants) | 7
  5-years post permanent restoration (Visit 14) | 3.4 (4.4)

6. Secondary Outcome: At Least One Surface With Plaque.
Description: Plaque was recorded as presence or absence of plaque by visual inspection on four surfaces at each implant site (mesially, distally, buccally and lingually).
Time Frame: as for outcome 5
Population: Intention to treat
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
Number analyzed (implants) | 62
implants
  Any plaque at permanent restoration (Visit 8) | 14
  Any plaque at 6-months post permanent restoration (Visit 9): number analyzed (implants) | 61
  Any plaque at 6-months post permanent restoration (Visit 9) | 32
  Any plaque at 1-year post permanent restoration (Visit 10): number analyzed (implants) | 61
  Any plaque at 1-year post permanent restoration (Visit 10) | 35
  Any plaque at 2-years post permanent restoration (Visit 11): number analyzed (implants) | 54
  Any plaque at 2-years post permanent restoration (Visit 11) | 28
  Any plaque at 3-years post permanent restoration (Visit 12): number analyzed (Participants) | 8
  Any plaque at 3-years post permanent restoration (Visit 12): number analyzed (implants) | 44
  Any plaque at 3-years post permanent restoration (Visit 12) | 35
  Any plaque at 5-years post permanent restoration (Visit 14): number analyzed (Participants) | 7
  Any plaque at 5-years post permanent restoration (Visit 14): number analyzed (implants) | 41
  Any plaque at 5-years post permanent restoration (Visit 14) | 23

7. Secondary Outcome: Any Bleeding on Implant (BoP)
Description: BoP was evaluated at each of the four surfaces around the implant site (mesially, distally, buccally and lingually), by using a periodontal probe. BoP was recorded as presence or absence of bleeding when probing to the bottom of the pocket.
Time Frame: as for outcome 5
Population: Intention to treat
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
Number analyzed (implants) | 62
implants
  Any surface with BoP at permanent restoration (Visit 8) | 24
  Any surface with BoP at 6-months post permanent restoration (Visit 9): number analyzed (implants) | 61
  Any surface with BoP at 6-months post permanent restoration (Visit 9) | 44
  Any surface with BoP at 1-year post permanent restoration (Visit 10): number analyzed (implants) | 61
  Any surface with BoP at 1-year post permanent restoration (Visit 10) | 39
  Any surface with BoP at 2-years post permanent restoration (Visit 11): number analyzed (implants) | 54
  Any surface with BoP at 2-years post permanent restoration (Visit 11) | 29
  Any surface with BoP at 3-years post permanent restoration (Visit 12): number analyzed (Participants) | 8
  Any surface with BoP at 3-years post permanent restoration (Visit 12): number analyzed (implants) | 44
  Any surface with BoP at 3-years post permanent restoration (Visit 12) | 29
  Any surface with BoP at 5-years post permanent restoration (Visit 14): number analyzed (Participants) | 7
  Any surface with BoP at 5-years post permanent restoration (Visit 14): number analyzed (implants) | 41
  Any surface with BoP at 5-years post permanent restoration (Visit 14) | 15

8. Secondary Outcome: Oral Health Impact Profile 14 (OHIP-14)
Description: Patient satisfaction was evaluated using the Oral Health Impact Profile 14 (OHIP-14). The questionnaire was filled in by the subjects before and after treatment with implants. OHIP-14 includes seven domains: functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. An example of an OHIP statement is "Have you had to interrupt meals because of problems with your teeth, mouth or dentures". Responses are based on a Likert scale (i.e., 0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, 4 = very often). The lowest possible total score (all question responses summed) of the OHIP-4 questionnaire is 0, and the highest possible score is 56. A high score is linked to a poor outcome.
Time Frame: At pre-surgical planning (Visit 2) on average 6 months before PR, and at 6-months after PR (Visit 9), at 1-year after PR (Visit 10), at 2-years after PR (Visit 11), at 3-years after PR (Visit 12), and at 5-years after PR (Visit 14).
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 12
units on a scale
  Overall (Q1-14) at pre-surgical planing (Visit 2) | 27.8 (16.13)
  Overall (Q1-14) at 6-months post permanent restoration: number analyzed (Participants) | 11
  Overall (Q1-14) at 6-months post permanent restoration | 5.2 (7.67)
  Overall (Q1-14) at 1-year post permanent restoration: number analyzed (Participants) | 11
  Overall (Q1-14) at 1-year post permanent restoration | 8.3 (10.85)
  Overall (Q1-14) at 2-years post permanent restoration: number analyzed (Participants) | 8
  Overall (Q1-14) at 2-years post permanent restoration | 4.5 (6.09)
  Overall (Q1-14) at 5-years post permanent restoration: number analyzed (Participants) | 7
  Overall (Q1-14) at 5-years post permanent restoration | 6.9 (8.84)

9. Secondary Outcome: Prosthetic Survival Rate on Subject Level
Description: A prosthetic restoration was considered a survived if the original restoration was still in place, regardless of its condition, at the follow-up visit.
Time Frame: At 1-year after PR (Visit 10), at 2-years after PR (Visit 11), at 3-years after PR (Visit 12), and at 5-years after PR (Visit 14).
Population: Intention to treat
Measure: Count of Units; unit: Prosthesis (Bridges)
Units Other Than Participants: Prosthesis (Bridges)
Arm/Group | ANKYLOS C/X Implant A 6.6
Number analyzed (Participants) | 11
Number analyzed (Prosthesis (Bridges)) | 11
Prosthesis (Bridges)
  At 1-year post permanent restoration: Original prosthesis still in place | 10
  At 1-year post permanent restoration: Original prosthesis not in place | 1
  At 2-years post permanent restoration: number analyzed (Participants) | 10
  At 2-years post permanent restoration: number analyzed (Prosthesis (Bridges)) | 10
  At 2-years post permanent restoration: Original prosthesis still in place | 10
  At 2-years post permanent restoration: Original prosthesis not in place | 0
  At 3-years post permanent restoration: number analyzed (Participants) | 8
  At 3-years post permanent restoration: number analyzed (Prosthesis (Bridges)) | 8
  At 3-years post permanent restoration: Original prosthesis still in place | 8
  At 3-years post permanent restoration: Original prosthesis not in place | 0
  At 5-years post permanent restoration: number analyzed (Participants) | 7
  At 5-years post permanent restoration: number analyzed (Prosthesis (Bridges)) | 7
  At 5-years post permanent restoration: Original prosthesis still in place | 7
  At 5-years post permanent restoration: Original prosthesis not in place | 0

ADVERSE EVENTS:
Time Frame: On average 5.5 years. Adverse event data were collected from enrollment (signing informed consent) up to study termination (Visit 14, 5 years after PR).
Description: Safety endpoints were Adverse Events (AE), Adverse Device Effects (ADE), Serious Adverse Events (SAE), Serious Adverse Device Effects (SADE) and Device Deficiencies (DD)
Arm/Group | ANKYLOS C/X Implant A 6.6
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANKYLOS C/X Implant A 6.6 (N=12)
Dental implant related event (Product Issues) | 8 (11)
Dental abutment related event (Product Issues) | 2 (2)
Dental prosthesis related event (Product Issues) | 2 (5)
Porcelain chipping (Product Issues) | 5 (10)
Peri-implant tissue related event (Investigations) | 4 (4)
Hypertension (Cardiac disorders) | 1 (1)
Hand infection (Infections and infestations) | 1 (1)
Back injury and spinal fusion surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Nickel allergy (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle spasm neck region (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar vertebrae surgery (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02656823/Prot_SAP_000.pdf